CLINICAL TRIAL: NCT04249037
Title: Prospective Pilot Study of the Efficacy, Safety and Tolerability of Bictegravir-Based HIV ART Same-Day Treatment Evaluations (B-HASTE)
Brief Title: Rapid Start vs. Standard Start Antiretroviral Therapy (ART) in HIV
Acronym: B-HASTE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: University of Colorado, Denver (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-0829
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — bictegravir; emtricitabine tenofovir alafenamide; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Rapid Start Group (Active Comparator): Same day antiretroviral therapy (ART) with bictegravir/emtricitabine/tenofovir alafenamide (BIC/F/TAF) + new diagnosis package with laboratory evaluations and social work referral.
  Interventions: Drug: bictegravir/emtricitabine/tenofovir alafenamide (BIC/F/TAF)
- Arm B: Standard Group (Placebo Comparator): Standard initiation of ART at the discretion of provider + new diagnosis package with laboratory evaluations and social work referral.
  Interventions: Drug: Standard initiation of antiretroviral therapy (ART)

INTERVENTIONS:
Drug: bictegravir/emtricitabine/tenofovir alafenamide (BIC/F/TAF) — A 30 day supply of Bictegravir 50mg/Emtricitabine 200mg/Tenofovir Alafenamide 25mg will be provided to the rapid start arm.
  Other Names: Biktarvy
  Arms: Arm A: Rapid Start Group
Drug: Standard initiation of antiretroviral therapy (ART) — Standard initiation of ART at the discretion of provider + new diagnosis package with laboratory evaluations and social work referral.
  Other Names: Standard of Care ART
  Arms: Arm B: Standard Group

SUMMARY:
This study plans to learn about whether starting HIV treatment very soon after diagnosis is more beneficial than waiting until entering routine clinical care after diagnosis.

DETAILED DESCRIPTION:
Randomized two arm, multi-site (three sites), open label pilot study conducted with laboratory evaluation and visits at entry, 4 weeks, 12 weeks, 24 weeks, 48 weeks and 96 weeks with laboratory evaluations and assessment if participants remain engaged in care.

Participants will be randomly assigned with equal probability to one of two arms:

Arm A: Same day antiretroviral therapy (ART) with bictegravir/emtricitabine/tenofovir alafenamide (BIC/F/TAF) + new diagnosis package with laboratory evaluations and social work referral.

Arm B: Standard initiation of ART at the discretion of provider + new diagnosis package with laboratory evaluations and social work referral.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 15 years and older in Colorado and 19 years and older in Nebraska. A waiver of parental consent is planned for individuals 15-17 in accordance with Colorado law which allows minors to consent for treatment for sexually transmitted infections, including HIV.
* Reactive HIV-1 on an approved fourth generation HIV-1 antibody/antigen test within 72 hours
* Any primary language with access to an interpreter by phone is included.

Exclusion Criteria:

* Pregnancy or intention to become pregnant in the next two years after enrollment
* Symptomatic acute HIV (with fever, rash, influenza-like symptoms)
* Creatinine clearance <30 mL/min by Cockcroft-Gault equation. (Therapy initiated will be terminated promptly in individuals who are found to have creatinine clearance <30 mL/min)
* Prior history of known HIV diagnosis
* Negative confirmatory HIV differentiation assays (therapy initiated will be terminated in individuals with negative tests and excluded from the primary analysis)
* Allergy to bictegravir, emtricitabine or tenofovir alafenamide
* Signs or symptoms of opportunistic infection with cryptococcal meningitis, tuberculosis or other infection that requires delay of initiation of antiretroviral therapy (up to the discretion of the site PI)
* Vulnerable populations including prisoners and individuals without decision making capacity
* Concommitant use of medications that are contraindicated with bictegravir, emtricitabine and tenofovir alafenamide including adefovir, carbamazepine, cladribine, dofetilide, fosphenytoin-phenytoin, oxcarbazepine, phenobarbital, primidone, rifampin, rifabutin, rifapentine, St. John's Wort, tipranavir

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Viral Suppression | 48 weeks
  Proportion of participants with viral suppression to <50 copies/mL at 48 weeks by FDA snapshot in the rapid-start ART arm compared to the standard of care arm.

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Dunlevy, MD, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Anschutz, Aurora, Colorado
  - University of Nebraska, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No